CLINICAL TRIAL: NCT05229822
Title: Prognostic Significance of Bacterial Translocation Markers as Predictors of Infectious and Inflammatory Complications in Acute Mechanical Bowel Obstruction
Brief Title: Bacterial Translocation Markers as Predictors of Infectious and Inflammatory Complications in Acute Bowel Obstruction
Status: Completed | Type: Observational
Sponsor: Karaganda Medical University (Other)
Collaborators: Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Sponsor
Other Study IDs: BT-ABO
Record Dates: First submitted 2022-01-21; First posted 2022-02-08 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Intestinal Obstruction; Colorectal Cancer; Post-Op Complication; Systemic Inflammatory Response Syndrome; Colon Tumor
Keywords: acute bowel obstruction; colon tumor; bacterial translocation; presepsin; lipopolysaccharide-binding protein; 16s rRNA; post-operative complications
MeSH Terms: conditions — Intestinal Obstruction; Colorectal Neoplasms; Postoperative Complications; Systemic Inflammatory Response Syndrome; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Malignant ABO: 60 patients with malignant acute bowel obstruction
  Interventions: Diagnostic Test: LBP; Diagnostic Test: sCD14-ST; Diagnostic Test: 16s rRNA
- CRC without ABO (control): 60 colorectal cancer patients without acute bowel obstruction (planned operations)
  Interventions: Diagnostic Test: LBP; Diagnostic Test: sCD14-ST; Diagnostic Test: 16s rRNA
- Benign ABO: 30 patients with benign acute bowel obstruction
  Interventions: Diagnostic Test: LBP; Diagnostic Test: sCD14-ST; Diagnostic Test: 16s rRNA

INTERVENTIONS:
Diagnostic Test: LBP — Determine any presence of LBP in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
Diagnostic Test: sCD14-ST — Determine any presence of sCD14-ST in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
Diagnostic Test: 16s rRNA — Determine any presence of 16s rRNA in mesenteric lymph nodes by PCR method.

SUMMARY:
Despite modern approaches to the diagnosis and treatment of acute bowel obstruction (ABO), postoperative mortality ranges from 5 to 32%, and complications occur up 23% of cases. One of the formidable infectious and inflammatory complications of ABO is sepsis. The main component of the development of sepsis in ABO is bacterial translocation (BT). BT is the migration of intestinal bacteria or their products through the intestinal mucosa into the mesenteric lymph nodes and further into normally sterile tissues and organs.

Today there are several methods for detecting BT:

1. direct method - the detection of 16s rRNA (ribosomal ribonucleic acid) in mesenteric lymph nodes (MLN);
2. indirect method - the detection of serum lipopolysaccharide-binding protein (LBP) and presepsin (Soluble CD14 subtype or sCD14-ST).

The aim of this study is to determine the diagnostic and prognostic significance of bacterial translocation as a predictor of the complications development in patients with malignant and benign acute bowel obstruction by assessing the relationship of biomarkers in the systemic circulation (LBP, sCD14-ST) with the detection of microorganism genes (16s rRNA) in mesenteric lymph nodes.

DETAILED DESCRIPTION:
For the early diagnosis of infectious and inflammatory complications, it is necessary to study LBP, sCD-14 and 16sRNA as bacterial translocation markers in patients with malignant and benign acute bowel obstruction, as well as in patients after planned surgical intervention for colon tumors. Based on changes in bacterial translocation biomarkers in the blood serum, it's suggested that patients with researched pathology can be stratified according to the risk level of developing infectious and inflammatory complications.

The study materials are blood serum and mesenteric lymph nodes (MLN). Venous blood sampling will be performed 1 hour before surgery, 24 and 72 hours after it. Venous blood will be collected in 5 ml vacutainers with a coagulation activator and a serum gel separator. It will be centrifuged for 20 minutes at 1000 x g, after which the gel completely separates the serum from the clot, forming a tight barrier.ELISA Kit for Lipopolysaccharide Binding Protein (LBP, Human) and for Presepsin (sCD14-ST, Human), from Cloud-Clone Corp. will be used to determine any presence of LBP and sCD14-ST. The analysis will be performed according to the manufacturer's instructions for an ELISA EVOLIS robotic system from BioRad.

The operating surgeon will perform a MLN sampling in sterile conditions during surgery after resection of the intestine from the mesentery of the gross specimen. MLN will be placed in a sterile tube without any fillers. The DNA will be extracted by the GeneJET Genomic DNA Purification Kit manufactured by Thermo Fisher Scientific, USA, in accordance with the manufacturer's instructions. The 16s rRNA bacteria in MLN will be detected by using real-time PCR and BIO-RAD CFX96 amplifier with 16s rRNA forward and reverse primers (U16SRT-F FACTCCTACGGGAGGGAGGCAGGT and U16SRT-R TATTACCGCGGCTGCTGGGC).

During the implementation, the resources of the Collective Use Laboratory of Research Center Non-profit Joint Stock Company (NJSC) "Karaganda Medical University" will be used.

This research is funded by the Science Committee of the Ministry of Education and Science of the Republic of Kazakhstan (Grant No. AP09260597).

ELIGIBILITY:
Inclusion Criteria:

* patients with malignant acute bowel obstruction,
* patients with benign acute bowel obstruction,
* colorectal cancer patients without acute bowel obstruction (planned operations).

Exclusion Criteria:

* age less than 18,
* pregnancy,
* patients with paralytic acute bowel obstruction,
* patients with HIV infection, liver cirrhosis,
* patient with an infectious process due to another pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant and benign acute bowel obstruction, colorectal cancer patients without acute bowel obstruction (planned operations) aged from 18, who are expected to undergo surgical treatment for this pathology.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yemek Turgunov, Pr., Study Chair — NJSC Karaganda Medical University; Alina Ogizbayeva, PhD student, Principal Investigator — NJSC Karaganda Medical University; Lyudmila Akhmaltdinova, PhD, Principal Investigator — NJSC Karaganda Medical University; Kairat Shakeyev, Pr., Principal Investigator — NJSC Karaganda Medical University; Dmitry Matyushko, PhD, Principal Investigator — Multidisciplinary hospital No. 1 of Karaganda; Miras Mugazov, PhD, Principal Investigator — NJSC Karaganda Medical University; Asylbek Zhumakaev, Master, Principal Investigator — Multidisciplinary hospital No. 3 of Karaganda; Irina Kadyrova, PhD, Principal Investigator — NJSC Karaganda Medical University
Locations (1):
- NJSC Karaganda Medical University, Karaganda, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gore RM, Silvers RI, Thakrar KH, Wenzke DR, Mehta UK, Newmark GM, Berlin JW. Bowel Obstruction. Radiol Clin North Am. 2015 Nov;53(6):1225-40. doi: 10.1016/j.rcl.2015.06.008. PMID 26526435
- [Background] Taylor MR, Lalani N. Adult small bowel obstruction. Acad Emerg Med. 2013 Jun;20(6):528-44. doi: 10.1111/acem.12150. PMID 23758299
- [Background] Roses RE, Folkert IW, Krouse RS. Malignant Bowel Obstruction: Reappraising the Value of Surgery. Surg Oncol Clin N Am. 2018 Oct;27(4):705-715. doi: 10.1016/j.soc.2018.05.010. Epub 2018 Jul 21. PMID 30213414
- [Background] Shwaartz C, Fields AC, Prigoff JG, Aalberg JJ, Divino CM. Should patients With obstructing colorectal cancer have proximal diversion? Am J Surg. 2017 Apr;213(4):742-747. doi: 10.1016/j.amjsurg.2016.08.005. Epub 2016 Sep 2. PMID 27742029
- [Background] Chiu HC, Lin YC, Hsieh HM, Chen HP, Wang HL, Wang JY. The impact of complications on prolonged length of hospital stay after resection in colorectal cancer: A retrospective study of Taiwanese patients. J Int Med Res. 2017 Apr;45(2):691-705. doi: 10.1177/0300060516684087. Epub 2017 Feb 7. PMID 28173723
- [Background] Simillis C, Kalakouti E, Afxentiou T, Kontovounisios C, Smith JJ, Cunningham D, Adamina M, Tekkis PP. Primary Tumor Resection in Patients with Incurable Localized or Metastatic Colorectal Cancer: A Systematic Review and Meta-analysis. World J Surg. 2019 Jul;43(7):1829-1840. doi: 10.1007/s00268-019-04984-2. PMID 30903246
- [Background] Wancata LM, Abdelsattar ZM, Suwanabol PA, Campbell DA Jr, Hendren S. Outcomes After Surgery for Benign and Malignant Small Bowel Obstruction. J Gastrointest Surg. 2017 Feb;21(2):363-371. doi: 10.1007/s11605-016-3307-8. Epub 2016 Oct 25. PMID 27783343
- [Background] Stubljar D, Skvarc M. Effective Strategies for Diagnosis of Systemic Inflammatory Response Syndrome (SIRS) due to Bacterial Infection in Surgical Patients. Infect Disord Drug Targets. 2015;15(1):53-6. doi: 10.2174/1871526515666150320161804. PMID 25809624
- [Background] Levy M, Kolodziejczyk AA, Thaiss CA, Elinav E. Dysbiosis and the immune system. Nat Rev Immunol. 2017 Apr;17(4):219-232. doi: 10.1038/nri.2017.7. Epub 2017 Mar 6. PMID 28260787
- [Background] Piton G, Capellier G. Biomarkers of gut barrier failure in the ICU. Curr Opin Crit Care. 2016 Apr;22(2):152-60. doi: 10.1097/MCC.0000000000000283. PMID 26808138
- [Background] Tsujimoto H, Ono S, Mochizuki H. Role of translocation of pathogen-associated molecular patterns in sepsis. Dig Surg. 2009;26(2):100-9. doi: 10.1159/000206143. Epub 2009 Mar 2. PMID 19252406
- [Background] MacFie J, Reddy BS, Gatt M, Jain PK, Sowdi R, Mitchell CJ. Bacterial translocation studied in 927 patients over 13 years. Br J Surg. 2006 Jan;93(1):87-93. doi: 10.1002/bjs.5184. PMID 16288452
- [Background] Fang L, Xu Z, Wang GS, Ji FY, Mei CX, Liu J, Wu GM. Directed evolution of an LBP/CD14 inhibitory peptide and its anti-endotoxin activity. PLoS One. 2014 Jul 15;9(7):e101406. doi: 10.1371/journal.pone.0101406. eCollection 2014. PMID 25025695
- [Background] Stehle JR Jr, Leng X, Kitzman DW, Nicklas BJ, Kritchevsky SB, High KP. Lipopolysaccharide-binding protein, a surrogate marker of microbial translocation, is associated with physical function in healthy older adults. J Gerontol A Biol Sci Med Sci. 2012 Nov;67(11):1212-8. doi: 10.1093/gerona/gls178. Epub 2012 Sep 7. PMID 22960476
- [Background] Kell DB, Pretorius E. On the translocation of bacteria and their lipopolysaccharides between blood and peripheral locations in chronic, inflammatory diseases: the central roles of LPS and LPS-induced cell death. Integr Biol (Camb). 2015 Nov;7(11):1339-77. doi: 10.1039/c5ib00158g. PMID 26345428
- [Background] Mussap M, Noto A, Fravega M, Fanos V. Soluble CD14 subtype presepsin (sCD14-ST) and lipopolysaccharide binding protein (LBP) in neonatal sepsis: new clinical and analytical perspectives for two old biomarkers. J Matern Fetal Neonatal Med. 2011 Oct;24 Suppl 2:12-4. doi: 10.3109/14767058.2011.601923. PMID 21740312
- [Background] van Maldeghem I, Nusman CM, Visser DH. Soluble CD14 subtype (sCD14-ST) as biomarker in neonatal early-onset sepsis and late-onset sepsis: a systematic review and meta-analysis. BMC Immunol. 2019 Jun 3;20(1):17. doi: 10.1186/s12865-019-0298-8. PMID 31159729
- [Background] Hosomi S, Yamagami H, Itani S, Yukawa T, Otani K, Nagami Y, Tanaka F, Taira K, Kamata N, Tanigawa T, Shiba M, Watanabe T, Fujiwara Y. Sepsis Markers Soluble IL-2 Receptor and Soluble CD14 Subtype as Potential Biomarkers for Complete Mucosal Healing in Patients With Inflammatory Bowel Disease. J Crohns Colitis. 2018 Jan 5;12(1):87-95. doi: 10.1093/ecco-jcc/jjx124. PMID 28961693
- [Background] Endo S, Suzuki Y, Takahashi G, Shozushima T, Ishikura H, Murai A, Nishida T, Irie Y, Miura M, Iguchi H, Fukui Y, Tanaka K, Nojima T, Okamura Y. Presepsin as a powerful monitoring tool for the prognosis and treatment of sepsis: a multicenter prospective study. J Infect Chemother. 2014 Jan;20(1):30-4. doi: 10.1016/j.jiac.2013.07.005. Epub 2013 Dec 11. PMID 24462421
- See also: Mierzchala M, Krzystek-Korpacka M, Gamian A, Durek G. Quantitative indices of dynamics in concentrations of lipopolysaccharide-binding protein (LBP) as prognostic factors in severe sepsis/septic shock patients - Comparison with CRP and procalcitonin / — http://doi.org/10.1016/j.clinbiochem.2011.01.012
- See also: Masson S, Caironi P, Fanizza C, Thomae R, Bernasconi R, Noto A, Oggioni R, Pasetti GS, Romero M, Tognoni G, Latini R, Gattinoni L. Circulating presepsin (soluble CD14 subtype) as a marker of host response in patients with severe sepsis or septic shock — https://doi.org/10.1007/s00134-014-3514-2

RESULTS

PARTICIPANT FLOW:
Groups:
- CRC Without ABO (Control): 60 colorectal cancer patients without acute bowel obstruction (planned operations)
  Lipopolysaccharide-binding protein (LBP): Determine any presence of LBP in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  soluble CD14 subtype (sCD14-ST): Determine any presence of sCD14-ST in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  16 subunits of ribosomal ribonucleic acid (16s rRNA): Determine any presence of 16s rRNA in mesenteric lymph nodes by PCR method.
- Malignant ABO: 60 patients with malignant acute bowel obstruction
  Lipopolysaccharide-binding protein (LBP): Determine any presence of LBP in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  soluble CD14 subtype (sCD14-ST): Determine any presence of sCD14-ST in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  16 subunits of ribosomal ribonucleic acid (16s rRNA): Determine any presence of 16s rRNA in mesenteric lymph nodes by PCR method.
- Benign ABO: 30 patients with benign acute bowel obstruction
  Lipopolysaccharide-binding protein (LBP): Determine any presence of LBP in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  soluble CD14 subtype (sCD14-ST): Determine any presence of sCD14-ST in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  16 subunits of ribosomal ribonucleic acid (16s rRNA): Determine any presence of 16s rRNA in mesenteric lymph nodes by PCR method.
Period: Overall Study
Arm/Group | CRC Without ABO (Control) | Malignant ABO | Benign ABO
Started | 60 | 60 | 30
Completed | 60 | 60 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The acceptance criteria are as follows: patients undergoing planned surgical intervention for colorectal tumor, patients with ABO of tumor and non-tumor genesis over 18 years of age.
  The exclusion criteria included: age under 18 years, pregnant women, patients with paralytic/dynamic ABO, patients with HIV infection, liver cirrhosis as well as those patients with an ongoing infectious process due to another pathology.
Groups:
- Malignant ABO: 60 patients with malignant acute bowel obstruction
  LBP: Determine any presence of LBP in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  sCD14-ST: Determine any presence of sCD14-ST in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  16s rRNA: Determine any presence of 16s rRNA in mesenteric lymph nodes by PCR method.
  TNM international classification of malignant neoplasm stages was used with grouping by stages I-IV according to the latest 8th revision of the classification.
- CRC Without ABO (Control): 60 colorectal cancer patients without acute bowel obstruction (planned operations)
  LBP: Determine any presence of LBP in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  sCD14-ST: Determine any presence of sCD14-ST in blood serum by ELISA method 1 hour before surgery, 24 and 72 hours after it.
  16s rRNA: Determine any presence of 16s rRNA in mesenteric lymph nodes by PCR method.
  TNM international classification of malignant neoplasm stages was used with grouping by stages I-IV according to the latest 8th revision of the classification.
- Total: Total of all reporting groups
Arm/Group | Malignant ABO | CRC Without ABO (Control) | Benign ABO | Total
Number analyzed (Participants) | 60 | 60 | 30 | 150
Age, Categorical [Count of Participants; unit: Participants] — Age was measured in complete years.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 26 | 26 | 20 | 72
    >=65 years | 34 | 34 | 10 | 78
Age, Continuous [Median (Inter-Quartile Range); unit: years] — For each group, the median age in years was calculated.
  years | 67.5 [58.5 to 78] | 66.5 [54 to 73] | 59.5 [43 to 70] | 66 [56 to 73.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 26 | 15 | 80
  Male | 21 | 34 | 15 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Region of Enrollment - four hospitals in the city of Karaganda, Kazakhstan: Regional Clinical Hospital, Professor H.J. Maqajanov Multidisciplinary Hospital, Multidisciplinary Hospital No. 1 of Karaganda city, Multidisciplinary Hospital No. 3 of Karaganda city
  participants
    Kazakhstan | 60 | 60 | 30 | 150
Stage of the tumor process [Count of Participants; unit: Participants] — Colon cancer is staged using the American Joint Committee on Cancer (AJCC) tumor/node/metastasis (TNM) classification and staging system (8th revision of the classification). In this system, I-IV stages are assigned on the basis of the characteristics of the primary tumor (T) and the extent of regional lymph node involvement (N) and distant metastasis (M). Stage IV was considered worse outcomes. Population: The stage of the tumor process (I-IV) is not applicable to the group "Benign ABO"
  Participants
    number analyzed (Participants) | 60 | 60 | 0 | 120
    I | 2 | 10 | 0 | 12
    II | 20 | 26 | 0 | 46
    III | 14 | 17 | 0 | 31
    IV | 24 | 7 | 0 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Participants With Post-operative Infectious and Inflammatory Complications
Description: Аny infectious and inflammatory complications in post-operative period (wound suppuration, anastomotic leak, аbdominal abscesses, peritonitis, sepsis, etc.)
Time Frame: Once (if any complication occurs during hospitalization - from 7 to 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Malignant ABO | CRC Without ABO (Control) | Benign ABO
Number analyzed (Participants) | 60 | 60 | 30
Participants
  - Post-operative infectious complications | 43 | 47 | 25
  + Post-operative infectious complications | 17 | 13 | 5

2. Secondary Outcome: LBP Level in Serum Blood
Description: LBP levels will be compared between groups/ subgroups and in each group/subgroup in dynamic.
Time Frame: 1 hour before surgery, 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Malignant ABO | CRC Without ABO (Control) | Benign ABO
Number analyzed (Participants) | 60 | 60 | 30
ng/mL
  LBP before surgery (ng/mL) | 1164.4 [826.4 to 1509.7] | 971.4 [816.9 to 1277.5] | 1015.1 [486.4 to 1543.3]
  LBP on the 3rd day after surgery (ng/mL) | 890.9 [703.2 to 1213.7] | 897.9 [712.5 to 1220.9] | 1180.0 [687.1 to 1392.3]

3. Secondary Outcome: sCD14-ST Level in Serum Blood
Description: sCD14-ST levels will be compared between groups/ subgroups and in each group/subgroup in dynamic.
Time Frame: 1 hour before surgery, 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Malignant ABO | CRC Without ABO (Control) | Benign ABO
Number analyzed (Participants) | 60 | 60 | 30
pg/mL
  sCD14-ST before surgery (pg/mL) | 571.7 [342.5 to 990] | 245.7 [167.9 to 403.4] | 485.2 [277.9 to 771.0]
  sCD14-ST on day 3 after surgery (pg/mL) | 527.8 [305.0 to 732.5] | 227.6 [163.5 to 419.8] | 386.5 [185.4 to 957.0]

4. Secondary Outcome: 16s rRNA in Mesenteric Lymph Nodes
Description: Presence or absence of 16s rRNA in mesenteric lymph nodes will be compared between groups/subgroups.
Time Frame: Once (MLN sampling in sterile conditions during surgery)
Measure: Number; unit: Count of Participants
Arm/Group | Malignant ABO | CRC Without ABO (Control) | Benign ABO
Number analyzed (Participants) | 60 | 60 | 5
Count of Participants
  Presence of 16s rRNA | 15 | 16 | 0
  Absence of 16s rRNA | 45 | 44 | 5

ADVERSE EVENTS:
Time Frame: During hospitalization (from 7 to 28 days)
Description: Not applicable. Because the study is observational, without any intervention
Arm/Group | Malignant ABO | CRC Without ABO (Control) | Benign ABO
All-Cause Mortality (participants affected / at risk) | 12/60 | 1/60 | 2/30
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/30
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT05229822/Prot_SAP_001.pdf